CLINICAL TRIAL: NCT02839655
Title: Prospective Study Assessing Thyroidectomy Using Robot
Acronym: EVATAR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-A00989-40; 2015/2273 (Other: CSET Number)
Record Dates: First submitted 2016-07-12; First posted 2016-07-21 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Patients With Thyroid Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Da Vinci Xi (Experimental)
  Interventions: Device: Da Vinci Xi

INTERVENTIONS:
Device: Da Vinci Xi

SUMMARY:
The robot-assisted surgery for benign and malignant thyroid tumors was widely developed in Asia and begins to spread in Western countries. The main advantage of the technique is to avoid a scar in the neck by placing it either in the axilla or at the hairline behind the ear to improve esthetic consequences and body image. It is not surgery minimally invasive but rather a way of remote access surgery.

Data from the literature including cohort studies and meta-analyzes attest the security of the procedure in comparison with classic thyroid surgery (which remains the "gold standard"). However there is few data on the effectiveness of the technique in terms of the completeness of the surgery, according to the routine standard criteria used in endocrinology and endocrine cancer, and no French medico-economic study has been performed.

ELIGIBILITY:
Inclusion Criteria:

1. Benign thyroid nodule or follicular or suspicious cytological (Bethesda classifications 2, 3, 4, or 5) requiring thyroid lobectomy or total thyroidectomy therapeutic or diagnostic
2. Differentiated thyroid cancers - CN0 (no suspicious lymph node in the central or lateral compartments on preoperative ultrasound - CN1A / b with lymph node metastases <or = 10 mm in areas VI, III and / or IV, detected on preoperative ultrasound - For which the indication of a lobectomy or total thyroidectomy, with or without dissection of the central compartment and / or lateral neck was put in multidisciplinary meeting
3. Patient with no cons-indication to thyroid surgery or without dissection
4. Patient general condition of WHO grade 0-1
5. Patient age > 18 years and able to comply with the protocol visits
6. Patient agreeing to undergo robot-assisted surgery, the incision being at patient choice, depending on the wishes concerning the location of the scar (Axillary or behind the ear channel)
7. Patient Information or his legal representative and signed consent enlightened
8. Patient affiliated to a system of social security or beneficiary of such a scheme

Exclusion Criteria:

1. A history of cervical surgery or external beam radiation therapy
2. Anomaly craniocervical hinge or symptomatic cervical spondylosis
3. Congenital or acquired shoulder or ipsilateral upper limb surgery (for axillary )
4. paralysis preoperatively ( a laryngoscopic examination will be performed systematically preoperatively )
5. tumors with obvious extra- thyroid extension or suspected during preoperative ( cT3T4 )
6. metastatic cervical lymphadenopathy > 10 mm during the preoperative
7. Pregnant women or during lactation
8. patient already included in another clinical trial with a molecule experimental

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Efficacy for benign tumor | Assessed 3 months after surgery
  If total thyroidectomy : rate of patients with thyroglobulin (Tg) under non- suppressive treatment with L-thyroxine ( LT4 ) <2 ng / ml to 3 months with a target value TSH between 0.5 and 2 ng / mL If lobectomy : size of the remaining thyroid ipsilateral to the surgery evaluated sonographically <11 mm ( larger diameter ) to 3 months
Efficacy for malignant tumor | Assessed 12 months after surgery
  Rate of patients in complete remission at 12 months, remission defined as no biological or radiological anomaly:
  * Tg / LT4 < 2 ng / ml in the absence of treatment with 131I ( in the absence of anti Tg antibodies) or Tg / LT4 <0.2 ng / mL in patients treated with 131I (absent anti Tg antibody )
  * Normal cervical ultrasound
  * Normal SPECT -CT if treatment with 131I
  * If realized : CT and / or normal 18 FDG - PET

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France

IPD SHARING:
Plan to Share IPD: No